CLINICAL TRIAL: NCT03603574
Title: A Randomized Comparison Between Epidural Waveform Analysis Through the Needle Versus the Catheter for Thoracic Epidural Blocks
Brief Title: Epidural Waveform Analysis for Thoracic Epidural Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Ramathibodi Hospital (Other); University of Chile (Other)
Responsible Party: Principal Investigator, De Tran, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-4669
Record Dates: First submitted 2018-06-25; First posted 2018-07-27 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Surgical Procedure, Unspecified
Keywords: Abdomen/surgery; Thoracic Surgery

STUDY DESIGN:
Intervention Model Description: Randomized trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessment will not be present during the performance of the epidural block and waveform analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EWA through the needle (Experimental): EWA through the needle group, 5 mL of normal saline are injected through the epidural needle after the occurrence of LOR. The needle is subsequently connected to the pressure transducer (leveled with the heart) via the sterile, rigid extension tubing. A satisfactory endpoint is defined as the presence of waveforms synchronized with arterial pulsations.
  Interventions: Device: EWA through the needle
- EWA through the catheter (Experimental): EWA through the catheter group, the epidural catheter is advanced 5 cm beyond the needle tip after the occurrence of LOR. Subsequently, the operator injects 5 mL of normal saline through the catheter and the latter is connected to the pressure transducer via the sterile, rigid extension tubing. A satisfactory endpoint is defined as the presence of waveforms synchronized with arterial pulsations.
  Interventions: Device: EWA through the catheter

INTERVENTIONS:
Device: EWA through the needle — In the EWA-N group, 5 mL of normal saline are injected through the epidural needle after the occurrence of loss-of-resistance (LOR). The needle is connected to the pressure transducer. A satisfactory endpoint is defined as the presence of waveforms synchronized with arterial pulsations. In the absence of pulsatile waveforms, the operator injects an additional 2.5 mL-bolus of normal saline through the epidural needle and reconnects the latter to the pressure transducer. If no waveforms are detected after the second injection, the operator removes the needle and reattempts the epidural block at a different intervertebral level. A maximum of 3 levels is permitted: if waveforms are still absent at the third level, the operator simply accepts LOR as the technical endpoint.
  Arms: EWA through the needle
Device: EWA through the catheter — In the EWA-C group, the epidural catheter is advanced 5 cm beyond the needle tip after the occurrence of LOR. Subsequently, the operator injects 5 mL of normal saline through the catheter and the latter is connected to the pressure transducer via the sterile, rigid extension tubing. A satisfactory endpoint is defined as the presence of waveforms. In the absence of pulsatile waveforms, the operator injects an additional 2.5 mL-bolus of saline through the catheter and reconnects the latter to the pressure transducer. If no waveforms are detected after the second injection are still absent at the third level, the operator simply accepts this position for catheter placement (intent-to-treat analysis).
  Arms: EWA through the catheter

SUMMARY:
Epidural waveform analysis (EWA) provides a simple confirmatory adjunct for loss-of-resistance (LOR): when the needle/catheter tip is correctly positioned inside the epidural space, pressure measurement results in a pulsatile waveform. Epidural waveform analysis can be carried out through the tip of the needle or the catheter. In this randomized trial, the objective is to compare epidural waveform analysis through the needle (EWA-N) and through the catheter (EWA-C) for thoracic epidural blocks.

DETAILED DESCRIPTION:
The epidural space is most commonly identified with loss-of-resistance (LOR). Though sensitive Epidural waveform analysis (EWA) provides a simple confirmatory adjunct for LOR. When the needle (or catheter) is correctly positioned inside the epidural space, pressure measurement at its tip results in a pulsatile waveform synchronized with arterial pulsations Currently, there exist two different methods for EWA. Since local anesthetic (LA) is administered through the catheter, pressure transduction through its tip ensures that it is properly positioned inside the epidural space prior to LA injection. Alternately, EWA can be performed through the needle prior to blind advancement of the epidural catheter.

Thus, in this randomized trial, the aim is to compare epidural waveform analysis through the needle (EWA-N) and through the catheter (EWA-C) for thoracic epidural blocks. The hypothesis is that, compared to EWA-C, EWA-N will result in a shorter performance time.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* American Society of Anesthesiologists classification 1-3
* body mass index between 20 and 35

Exclusion Criteria:

* adults who are unable to give their own consent
* coagulopathy
* renal failure
* hepatic failure
* allergy to local anesthetic
* pregnancy
* prior surgery in the thoracic spine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
Performance time of block | From skin infiltration until local anesthetic administration through the needle or catheter, up to 60 minutes
  temporal interval in minutes between skin infiltration and local anesthetic administration through the epidural catheter (after obtaining a satisfactory waveform either through the needle or through the catheter depending on randomized group assignment).

SECONDARY OUTCOMES:
Incidence of successful epidural block | 15 minutes after the administration of local anesthetic through the epidural catheter
  bilateral block to ice in at least 2 dermatomes
Procedural pain during epidural block assessed by the numeric rating scale | From the performance of the epidural block until induction of general anesthesia, up to 2 hours
  pain in the back of the patient, related to the performance of the epidural block, using a numeric rating scale from 0 to 10 points (0=no pain and 10= worst imaginable pain)
Postoperative pain related to surgical incision assessed by the numeric rating scale | twice a day from the arrival at PACU or until catheter removal, up to 5 days
  pain at rest and upon deep breathing/coughing, measured using a numeric rating scale from 0 to 10 points ((0=no pain and 10= worst imaginable pain)
Local anesthetic consumption | once a day from the arrival at PACU or until catheter removal, up to 5 days
  amount of local anesthetic consumed
Breakthrough opioid consumption (if required) | once a day from the arrival at PACU or until catheter removal, up to 5 days
  amount of opioids consumed
Incidence of adverse events | Once a day from catheter insertion until removal, up to 5 days
  side effects related to the performance of the epidural block (eg, dural/vascular puncture, paresthesia) or breakthrough opioids (nausea, vomiting, pruritus, somnolence, respiratory depression)

CONTACTS AND LOCATIONS:
Overall Officials: De Q Tran, MD, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Hospital Clínico Universidad de Chile, Santiago, RM, Chile
- Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran DQ, Gonzalez AP, Bernucci F, Finlayson RJ. Confirmation of loss-of-resistance for epidural analgesia. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):166-73. doi: 10.1097/AAP.0000000000000217. No abstract available. PMID 25642911
- [Background] Sharrock NE. Recordings of, and an anatomical explanation for, false positive loss of resistance during lumbar extradural analgesia. Br J Anaesth. 1979 Mar;51(3):253-8. doi: 10.1093/bja/51.3.253. PMID 435350
- [Background] BONICA J. Continuous peridural block. Anesthesiology. 1956 Jul-Aug;17(4):626-30. No abstract available. PMID 13327296
- [Background] Lirk P, Kolbitsch C, Putz G, Colvin J, Colvin HP, Lorenz I, Keller C, Kirchmair L, Rieder J, Moriggl B. Cervical and high thoracic ligamentum flavum frequently fails to fuse in the midline. Anesthesiology. 2003 Dec;99(6):1387-90. doi: 10.1097/00000542-200312000-00023. PMID 14639154
- [Background] Lirk P, Moriggl B, Colvin J, Keller C, Kirchmair L, Rieder J, Kolbitsch C. The incidence of lumbar ligamentum flavum midline gaps. Anesth Analg. 2004 Apr;98(4):1178-1180. doi: 10.1213/01.ANE.0000101486.41355.35. PMID 15041621
- [Background] Chayen D, Nathan H, Chayen M. The psoas compartment block. Anesthesiology. 1976 Jul;45(1):95-9. doi: 10.1097/00000542-197607000-00019. No abstract available. PMID 937760
- [Background] Eason MJ, Wyatt R. Paravertebral thoracic block-a reappraisal. Anaesthesia. 1979 Jul-Aug;34(7):638-42. doi: 10.1111/j.1365-2044.1979.tb06363.x. PMID 517716
- [Background] Leurcharusmee P, Arnuntasupakul V, Chora De La Garza D, Vijitpavan A, Ah-Kye S, Saelao A, Tiyaprasertkul W, Finlayson RJ, Tran DQ. Reliability of Waveform Analysis as an Adjunct to Loss of Resistance for Thoracic Epidural Blocks. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):694-7. doi: 10.1097/AAP.0000000000000313. PMID 26469364
- [Background] Tran DQ, Van Zundert TC, Aliste J, Engsusophon P, Finlayson RJ. Primary Failure of Thoracic Epidural Analgesia in Training Centers: The Invisible Elephant? Reg Anesth Pain Med. 2016 May-Jun;41(3):309-13. doi: 10.1097/AAP.0000000000000394. PMID 27035462
- [Background] Arnuntasupakul V, Van Zundert TC, Vijitpavan A, Aliste J, Engsusophon P, Leurcharusmee P, Ah-Kye S, Finlayson RJ, Tran DQ. A Randomized Comparison Between Conventional and Waveform-Confirmed Loss of Resistance for Thoracic Epidural Blocks. Reg Anesth Pain Med. 2016 May-Jun;41(3):368-73. doi: 10.1097/AAP.0000000000000369. PMID 26894628
- [Background] de Medicis E, Tetrault JP, Martin R, Robichaud R, Laroche L. A prospective comparative study of two indirect methods for confirming the localization of an epidural catheter for postoperative analgesia. Anesth Analg. 2005 Dec;101(6):1830-1833. doi: 10.1213/01.ANE.0000184130.73634.BE. PMID 16301268
- [Background] de Medicis E, Pelletier J, Martin R, Loignon MJ, Tetrault JP, Laroche L. Technical report: optimal quantity of saline for epidural pressure waveform analysis. Can J Anaesth. 2007 Oct;54(10):818-21. doi: 10.1007/BF03021709. PMID 17934163
- [Derived] Tangjitbampenbun A, Layera S, Arnuntasupakul V, Apinyachon W, Venegas K, Godoy J, Aliste J, Bravo D, Blanch A, Webar J, Saadawi M, Owen A, Finlayson RJ, Tran DQ. Randomized comparison between epidural waveform analysis through the needle versus the catheter for thoracic epidural blocks. Reg Anesth Pain Med. 2019 May 14:rapm-2019-100478. doi: 10.1136/rapm-2019-100478. Online ahead of print. PMID 31092706